CLINICAL TRIAL: NCT00318253
Title: The Effects of Cranberry Juice on Urine and Bacterial Adhesion to Cells
Brief Title: The Effects of Cranberry Juice on Bacterial Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Dr. G. Reid, Lawson Health Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: R-06-704; SP 0732
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Bacterial Vaginosis; Oxaluria
Keywords: Cranberry juice; Antiadhesion; Urinary tract infection; vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial; Hyperoxaluria; Urinary Tract Infections; Vaginal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cranberry juice

SUMMARY:
The study is based on the hypothesis that consumption of cranberry juice products results in the production of metabolites in the urine that have anti-adhesive properties on bacteria. A crossover study using 12 healthy women will be given different cranberry products or water as a control and their urine will be analyzed for anti-adhesive effects and compared to the properties of the urine. Cranberry juice will also be evaluated for its effect on vaginal microflora.

DETAILED DESCRIPTION:
Hypothesis: Metabolites in cranberry juice, have anti-adhesive properties for uropathogenic bacteria but they do not disturb the normal vaginal flora.

Study design and assays:

A crossover study design using 12 healthy women will be conducted for 50 days. The anti-adhesive properties of the urine will be determined using uropathogens and changes in the vaginal microflora will be evaluated.

Participants:

The subjects will be healthy premenopausal women aged 19-45, who have no history of chronic urinary tract infection or have had a urinary tract infection in the past 12 months, and are currently not taking antibiotics or any supplements to prevent UTI, including cranberry juice. The subjects must not have urinary tract abnormalities, requiring catheterization for micturition, be pregnant, or diabetic or have allergies to berry juices. Each test phase is 1 week (7 days) and the following protocol will be followed:

Subjects 1-3 Test phase I: water; washout phase Test phase II: cranberries; washout phase Test phase III: cranberry juice- 1/day; washout phase Test phase IV: cranberry juice- 2/day

4-6 Test phase I: cranberry juice- 2/day; washout phase Test phase II: water; washout phase Test phase III: cranberries; washout phase Test phase IV: cranberry juice- 1/day

7-9 Test phase I: cranberry juice- 1/day; washout phase Test phase II: cranberry juice- 2/day; washout phase Test phase III: water; washout phase Test phase IV: cranberries

10-12 Test phase I: cranberries; washout phase Test phase II: cranberry juice- 1/day; washout phase Test phase III: cranberry juice- 2/day; washout phase Test phase IV: water

During the washout period, the subjects will return to their normal diet with no added beverage or food, although again no cranberry juice can be consumed. The beverages/food to be taken for the 7 day phases comprise:

1. Water - Control group
2. Cranberry juice 1/day
3. Cranberry juice 2/day
4. Cranberries (dried)

Regime and sampling:

A mid stream urine sample will be collected to evaluate the anti-adhesive effects of the various treatments.

Mid stream urine will also be collected to evaluate anti-adhesive properties of the urine, and determine if changes occur following washout.

A 24 h urine will be collected after 3-4 days of each phase for urinalysis.

Vaginal swabs will be collected to determine the effect, if any, of the foods on the composition of the vaginal microflora.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-45 years
* Healthy pre-menopausal female volunteers with no history of urinary tract infections over the past 12 months.

Exclusion Criteria:

* Experienced a urinary tract infection in the past 12 months
* Receiving antibiotic therapy or supplements to prevent urinary tract infections
* Pregnant, postmenopausal or outside of the age range (19-45 years old)
* Anatomical abnormality of the urinary tract, such as following surgery
* Using a catheter to manage micturition
* Diabetic
* Allergic to berry juices

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
bacterial adhesion to tissue cells
microbial population shifts in vaginal tract

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, MBA, Principal Investigator — The Lawson Health Research Institute and The University of Western Ontario